CLINICAL TRIAL: NCT02789982
Title: Using Reconsolidation Blockade to Treat Trauma Related Disorders After Paris Attacks: an Effectiveness Study
Acronym: PARIS-MEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P151201; 2016-000257-12 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-06-03 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; Trauma related disorders; Reconsolidation blockade; Paris attacks
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reconsolidation blockade (Experimental): β-adrenergic blocker propranolol 1 mg / kg to each of the 6 treatment sessions
  Interventions: Drug: β-adrenergic blocker propranolol
- Treatment as usual (Active Comparator): Treatment as usual like SSRIs, psychotherapy, ...
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Drug: β-adrenergic blocker propranolol
  Arms: Reconsolidation blockade
Behavioral: Treatment as usual
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is: (1) to examine the effectiveness of reconsolidation blockade as a treatment for trauma-related disorders, (2) to evaluate the feasibility of implementing this new treatment on a large scale in a short delay. This clinical trial as been set up in response to the Paris attacks to increase treatment capacity of the AP-HP (Assistance Publique des Hopitaux de Paris) hospital network.. Reconsolidation blockade will be compared to treatment as usual (TAU), on symptoms reduction after 6 weeks of treatment. In order to measure effectiveness and cost-utility, socioeconomic measures, quality of life and social functioning outcomes will be measured pre- and post-treatment as well as 3 and 12 months after study enrollment.

DETAILED DESCRIPTION:
The November 13th Paris attacks were the most violent and devastating events to occur in France since World War II. A large number of persons are likely to develop PTSD or trauma-related disorders, especially victims directly involved, their families, as well as the the first responders. In this context, there is an urgent need to enhance treatment resources. Psychotherapy is known to be effective but it is costly, and require qualified professionals. Pharmacotherapy (e.g., selective serotonin reuptake inhibitor,SSRIs) is also considered effective. However, side effects often lead patients to abandon their treatment. An alternative evidence-based intervention is the use of the β-adrenergic blocker propranolol used to interfere with the reconsolidation of a recalled traumatic memory, so as to reduce its strength over time. This clinical trial will evaluate the effectiveness and cost-utility of reconsolidation blockade compared to treatment as usual. The study involves four assessments: pre- and post-treatment and 13 weeks and 1 year follow up. The outcome measures include: PTSD symptoms, socioeconomic variables, quality of life and social functioning measures. The investigators hypothesize that all patients will improve. However, patients receiving reconsolidation blockade will recover faster than treatment as usual. Finally, investigators hypothesize that reconsolidation blockade will be well accepted both by the professionals and the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Suffer from PTSD, adjustment disorders or other specified trauma- and stressor-related disorder
* PTSD Checklist - Specific (PCL-S) > 44
* Clinical Global Impression (CGI) > 3
* Informed Consent Form signed
* Fluency in French

Exclusion Criteria:

Reconsolidation blockade group:

* Resting systolic blood pressure < 100 mm Hg
* Resting heart rate < 55 beats per minute
* EKG significantly abnormal
* Medical contraindication to use propranolol
* Current use of medication that involve potentially dangerous interactions with propranolol
* Previous adverse reaction to a β-adrenergic blocker
* Current use of a β-adrenergic blocker
* Patients taking psychotropic drugs which may interact with propranolol will be examined on a case-by-case basis

Both groups:

* Subject under legal protection
* Bipolar or psychotic disorder
* Head trauma for less than one year or with clinical symptoms and neurological sequelae
* Proven severe suicide risk (Mini-S and clinical assessment)
* Opioid addiction or current alcohol dependence
* Patients using SSRI for less than 2 months
* Absence of affiliation to National french social security system
* Pregnant or breastfeeding woman or without effective contraception

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The PTSD Checklist (PCL-S) | change from baseline to 12 months follow-up
  The PCL-S is a 17-item self-report scale assessing DSM-IV-TR PTSD symptoms in the past week from the perspective of the patient. The PSL-S range between 17 (no symptom) and 85 (maximum score)
Medical resources use | from baseline to 12 months follow-up
  Costs, in Euros, related to healthcare utilization and work status are evaluated with the MEDico-Economic Questionnaire (MEDEC) adapted from the Client Service Receipt Inventory in order to meet the specificity of the French Health system
Quality of life assessed by EQ-5D-5L Euroquol questionnaire | at 12- months follow-up
  The EQ-5D-5L assesses five health dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated on five levels of severity. The levels of severity for each dimension ranges from no problems (1) to extreme problems/unable to perform (0)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno MILLET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (20):
- France (19):
  - Hôpital Albert Chenevier, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Corentin Celton, Issy-les-Moulineaux
  - Grand Hôpital EST FRANCILIEN - site de Marne-la-Vallée, Jossigny
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU et CIC de LILLE, Lille
  - Grand Hôpital EST FRANCILIEN - site de Meaux, Meaux
  - Chu Pasteur, Nice
  - Centre Hospitalier Sainte Marie, Nice
  - Hôpital Maison Blanche Hauteville, Paris
  - Hôpital Saint Antoine, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Tenon, Paris
  - Hôpital Sainte-Anne, Paris
  - Centre Hospitalier Henri Laborit, Poitiers
  - EPS Ville Evrard - site de Saint Denis, Saint-Denis
  - Hôpitaux de Saint Maurice, Saint-Maurice
  - Centre Hospitalier du Rouvray, Sotteville-lès-Rouen
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request :
  The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Mallet C, Chick CF, Maatoug R, Fossati P, Brunet A, Millet B. Memory reconsolidation impairment using the beta-adrenergic receptor blocker propranolol reduces nightmare severity in patients with posttraumatic stress disorder: a preliminary study. J Clin Sleep Med. 2022 Jul 1;18(7):1847-1855. doi: 10.5664/jcsm.10010. PMID 35404227
- [Derived] Brunet A, Ayrolles A, Gambotti L, Maatoug R, Estellat C, Descamps M, Girault N, Kalalou K, Abgrall G, Ducrocq F, Vaiva G, Jaafari N, Krebs MO, Castaigne E, Hanafy I, Benoit M, Mouchabac S, Cabie MC, Guillin O, Hodeib F, Durand-Zaleski I, Millet B. Paris MEM: a study protocol for an effectiveness and efficiency trial on the treatment of traumatic stress in France after the 2015-16 terrorist attacks. BMC Psychiatry. 2019 Nov 8;19(1):351. doi: 10.1186/s12888-019-2283-4. PMID 31703570